CLINICAL TRIAL: NCT02853773
Title: Acute Effects of Artificial Sweeteners and Sugar on the Brain Dynamics to Food Image Viewing. An Exploratory, Monocentric, Randomized Controlled Trial in Healthy Young Men
Brief Title: Effects of Consuming Artificial Sweeteners and Sugar on Cerebral and Physiological Responses
Acronym: SUGART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Full professor, University of Lausanne
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 353/15
Record Dates: First submitted 2016-02-08; First posted 2016-08-03 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-07

CONDITIONS: Normal Subjects
Keywords: sweeteners; sugar; EEG; food viewing; food intake
MeSH Terms: interventions — Sweetening Agents; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Artificial sweetener (Experimental): Effects of co-ingestion of artificially sweetened beverage on the response to a test meal
  Interventions: Other: ingestion of a test meal with sweetener
- Sugar (Active Comparator): Effects of co-ingestion of sugar-sweetened beverage on the response to a test meal
  Interventions: Other: ingestion of a test meal with sweetener
- Water (Active Comparator): Effects of co-ingestion of water on the response to a test meal
  Interventions: Other: ingestion of a test meal with water

INTERVENTIONS:
Other: ingestion of a test meal with sweetener — participants will ingest a test meal containing 55% carbohydrate, 30% fat and 15% protein with artificially sweetened drinks
  Arms: Artificial sweetener
Other: ingestion of a test meal with sweetener — participants will ingest a test meal containing 55% carbohydrate, 30% fat and 15% protein with sugary drinks drinks
  Arms: Sugar
Other: ingestion of a test meal with water — participants will ingest a test meal containing 55% carbohydrate, 30% fat and 15% protein with waters
  Arms: Water

SUMMARY:
This study aims at investigating the acute influence of artificially sweetened beverages consumption (as compared with sugar-sweetened beverages and water consumption) on brain responses to the viewing of food images, on physiological responses (gut-derived hormones and lipid metabolites) and on the food intake behavior.

DETAILED DESCRIPTION:
This study is made on a randomized controlled crossover design including three conditions (water, sugar, artificial sweeteners). Measurements will be performed in fasting and fed conditions. The test-meal will comprise either an artificially or sugar-sweetened beverage or water (control). The spatio-temporal brain dynamics to the viewing of food pictures will be assessed by means of electroencephalography (EEG) recordings and electrical neuroimaging analyses. Venous blood and urine will be collected. Blood pressure, cardiac frequency and bio-impedance measurements will be performed. Food intake behavior will be assessed by means of questionnaires and a free-choice buffet. Each tested condition (water, sugar, artificial sweeteners) will be preceded by a run-in period during which the participants' diet will be controlled (2-day isoenergetic diet).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Caucasian
* Right-handed
* Weak to normal physical activity (< 3hours per week)
* Normal-weight (19<BMI<25 kg/m2)
* Regular consumption of sugar-sweetened beverages (>33cl per week)

Exclusion Criteria:

* Consumption of artificially sweetened beverages exceeding 33cl per week
* Diabetes
* Cardiovascular, kidney, hepatic and/or psychological disorders
* Blood pressure at rest > 140/90mmHg
* Body weight < 50kg
* Hemoglobin < 13.5g/dl
* Ferritin < 50microg/l
* Drug consumption
* Alcohol consumption (>10g/day)
* Smoking
* Any particular diet (e.g. vegetarianism), food allergy and/or intolerance
* Body weight gain or loss of >3kg during the last 3 months

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Spatio-temporal brain dynamics | differences observed between 60 min before and 60 min after ingestion of a test meal
  Spatio-temporal brain dynamics to the viewing of food will be assessed by means of electroencephalography recordings.

SECONDARY OUTCOMES:
Changes in concentration of blood insulin | -120 min before ingestion of a test meal, and 30, 60, 90, 150, and 210 min after ingestion of a test meal
  Blood substrate concentration will be measured in fasting conditions and after ingestion of a test meal
Changes in concentration of blood triglyceride | -120 min before ingestion of a test meal, and 30, 60, 90, 150, and 210 min after ingestion of a test meal
  Blood substrate concentration will be measured in fasting conditions and after ingestion of a test meal
Changes in concentration of blood Fibroblast Growth Factor (FGF)-21 | -120 min before ingestion of a test meal, and 30, 60, 90, 150, and 210 min after ingestion of a test meal
  Blood substrate concentration will be measured in fasting conditions and after ingestion of a test meal
spontaneous food intake | 240 min after ingestion of a test meal
  Food intake behavior will be assessed by monitoring spontaneous food intake when offered a free-choice buffet.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, Professor, Principal Investigator — Department of Physiology, University of Lausanne, Switzerland
Locations (1):
- Department of Physiology, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No